CLINICAL TRIAL: NCT00111605
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of an HIV-1 Gag DNA Vaccine With or Without IL-12 DNA Adjuvant, Boosted With Homologous Plasmids in Healthy, HIV-1 Uninfected Adult Participants
Brief Title: Study of an HIV Preventive Vaccine Given With or Without an Adjuvant in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 060; 10057 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2005-05-23; First posted 2005-05-24 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: AIDS Vaccines; HIV Vaccines; HIV Preventive Vaccine; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (7):
- 1 (Experimental): HIV gag DNA vaccine or placebo on Days 0, 28, and 84
  Interventions: Biological: HIV-1 gag DNA; Biological: Sodium chloride injection (0.9%)
- 2 (Experimental): HIV gag DNA vaccine plus 100 mcg of IL-12 or placebo on Days 0, 28, and 84
  Interventions: Biological: HIV-1 gag DNA; Biological: HIV-1 gag DNA plus IL-12 DNA adjuvant; Biological: Sodium chloride injection (0.9%)
- 3 (Experimental): HIV gag DNA vaccine plus 500 mcg of IL-12 or placebo on Days 0, 28, and 84
  Interventions: Biological: HIV-1 gag DNA; Biological: HIV-1 gag DNA plus IL-12 DNA adjuvant; Biological: Sodium chloride injection (0.9%)
- 4 (Experimental): HIV gag DNA vaccine plus 1,500 mcg of IL-12 or placebo on Days 0, 28, and 84
  Interventions: Biological: HIV-1 gag DNA; Biological: HIV-1 gag DNA plus IL-12 DNA adjuvant; Biological: Sodium chloride injection (0.9%)
- 5 (Experimental): HIV gag DNA vaccine or placebo on Days 0, 28, 84, 168, and 273
  Interventions: Biological: HIV-1 gag DNA; Biological: Sodium chloride injection (0.9%)
- 6 (Experimental): HIV gag DNA vaccine plus IL-12 or placebo on Days 0, 28, and 84 plus CTL MEP/RC529-SE/GM-SCF booster vaccine on Days 168 and 273
  Interventions: Biological: HIV-1 gag DNA; Biological: HIV-1 gag DNA plus IL-12 DNA adjuvant; Biological: CTL MEP/RC529-SE/GM-CSF (CTL MEP vaccine); Biological: Sodium chloride injection (0.9%)
- 7 (Experimental): HIV gag DNA vaccine plus IL-12 DNA adjuvant or placebo on Days 0 and 84
  Interventions: Biological: HIV-1 gag DNA; Biological: Sodium chloride injection (0.9%)

INTERVENTIONS:
Biological: HIV-1 gag DNA — A 0.75 mL intramuscular injection of HIV gag DNA vaccine into the deltoid
Biological: HIV-1 gag DNA plus IL-12 DNA adjuvant — Injection IL-12 DNA adjuvant intramuscularly into the deltoid
  Arms: 2; 3; 4; 6
Biological: CTL MEP/RC529-SE/GM-CSF (CTL MEP vaccine) — A 1 mL intramuscular injection in the deltoid
  Arms: 6
Biological: Sodium chloride injection (0.9%) — All placebo groups will receive an intramuscular injection of sodium chloride (0.9%) in the deltoid.
  Group 1 will receive a 0.75 mL injection on Days 0, 28, and 84. Group 2 will receive a 0.8 mL injection on Days 0, 28, and 84. Group 3 will receive a 1.0 mL injection on Days 0, 28, and 84. Group 4 will receive a 1.5 mL injection on Days 0, 28, and 84. Group 5 will receive a 0.75 mL injection on Days 0, 28, 84, 168, and 273. Group 6 will receive a 1.5 mL injection on Days 0, 28, 84, 168, and 273. Group 7 will receive a 1.5 mL injection on Days 0, 28, and 84 and a 1 mL injection into the deltoid on Days 168 and 273.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of an experimental HIV vaccine. The vaccine will be given with or without IL-12 DNA adjuvant (at three escalating doses of 100, 500, and 1,500 mcg respectively), a substance that helps the body respond to a vaccine. This study will also determine the safety and tolerability of an experimental HIV vaccine boosted with two adjuvants.

DETAILED DESCRIPTION:
The HIV epidemic is a major global health challenge, causing tremendous human suffering and economic loss throughout the world. The need for a safe, effective, and affordable HIV preventive vaccine is critical. This study will determine the safety and immunogenicity of an experimental HIV vaccine, HIV-1 gag DNA, given with or without an IL-12 adjuvant and boosted HIV-1 gag DNA with or without IL-12 DNA adjuvant.

This study will comprise two parts (Parts A and B). Part A will last 9 months and Part B, 15 months. Part A will consist of 48 participants enrolled in 4 groups. Group 1 participants will be randomly assigned to receive the gag DNA vaccine or placebo. Participants in Groups 2, 3, and 4 will be randomly assigned to receive the gag DNA vaccine and either 100 mcg, 500 mcg, or 1,500 mcg IL-12 DNA or placebo. Vaccinations for Groups 1 through 4 will be given intramuscularly and will occur at study entry and at Months 1 and 3.

Part B will consist of 96 participants, enrolled in 3 groups. Participants in Part B will receive their first vaccination 2 weeks after Part A participants receive their second vaccination. Group 5 participants will receive either the HIV-1 gag DNA vaccine or placebo. Group 6 participants will receive either the HIV-1 gag DNA vaccine plus IL-12 DNA or placebo. Vaccinations for Groups 5 and 6 will occur at study entry and at Months 1, 3, 6, and 9. Group 7 participants will receive either the gag DNA vaccine plus IL-12 DNA or placebo at study entry and at Months 1 and 3. Throughout the study, blood and urine collections will occur, physical exams will be conducted, HIV testing and counseling will be offered, and interviews and questionnaires will be completed.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Access to a participating HIV Vaccine Trials Unit (HVTU)
* Willing to receive HIV test results
* Willing and able to comply with all study requirements
* In good general health
* Willing to use acceptable methods of contraception for at least 21 days prior to study entry and until the last study visit. More information about this criterion can be found in the protocol.
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (anti-HCV) antibody negative or negative HCV PCR if anti-HCV antibody is positive
* Weighs of or greater than 110 pounds (50 kg)

Exclusion Criteria:

* HIV infection
* HIV vaccines or placebos in prior HIV trial
* Immunosuppressive medications within 168 days prior to first study vaccination
* Blood products within 120 days prior to first study vaccination
* Live attenuated vaccines within 30 days prior to first study vaccination
* Medically indicated subunit or killed vaccines within 14 days prior to first study vaccination
* Pneumococcal vaccine within 14 days prior to first study vaccination
* Allergy treatment with antigen injections within 30 days prior to first study vaccination
* Current anti-tuberculosis (TB) preventive therapy or treatment
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health
* Any medical, psychiatric, or social condition that would interfere with the study. More information about this criterion can be found in the protocol.
* Any job-related responsibility that would interfere with the study
* Allergies to local amide-type anesthetics
* Serious adverse reactions to vaccines, including hypersensitivity and related symptoms. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection. Participants who have been fully treated for syphilis over 6 months prior to study entry are not excluded.
* Moderate to severe asthma. More information on this criterion can be found in the protocol.
* Type 1 or type 2 diabetes mellitus. Participants with histories of isolated gestational diabetes are not excluded.
* Thyroid disease or surgical removal of the thyroid requiring medication during the 12 months prior to study entry
* Accumulation of fluid in the blood vessels (angioedema) within 3 years prior to study entry, with episodes requiring medication in the 2 years prior to study entry
* Hypertension that is not well controlled by medication OR blood pressure of 150/100 or higher at study entry
* Body mass index (BMI) of 40 or greater OR BMI of 35 or greater, if certain criteria are met. More information about these criteria can be found in the protocol.
* Bleeding disorder
* Cancer. Participants with surgically removed cancer that, in the opinion of the investigator, is unlikely to recur are not excluded.
* Absence of the spleen
* Plans to become pregnant during the study
* Pregnancy or breastfeeding

Exclusion Criterion for Participants in Part B:

* Allergies to yeast-derived products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Safety, as judged by local and systemic reactogenicity signs and symptoms, laboratory measures of safety, and adverse and serious experiences | Throughout the study

SECONDARY OUTCOMES:
Immunogenicity, as judged by HIV-specific cellular responses assessed by interferon-gamma ELISpot assays and by intracellular cytokine staining (ICS) | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Spyros Kalams, MD, Study Chair — Vanderbilt University; Scott Parker, MD, Study Chair — University of Alabama at Birmingham
Locations (4):
- United States (3):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
- Chiang Mai Univ. HVTN CRS, Chiang Mai, Thailand

REFERENCES:
- [Background] Bolesta E, Gzyl J, Wierzbicki A, Kmieciak D, Kowalczyk A, Kaneko Y, Srinivasan A, Kozbor D. Clustered epitopes within the Gag-Pol fusion protein DNA vaccine enhance immune responses and protection against challenge with recombinant vaccinia viruses expressing HIV-1 Gag and Pol antigens. Virology. 2005 Feb 20;332(2):467-79. doi: 10.1016/j.virol.2004.09.043. PMID 15680412
- [Background] Letvin NL. Progress toward an HIV vaccine. Annu Rev Med. 2005;56:213-23. doi: 10.1146/annurev.med.54.101601.152349. PMID 15660510
- [Background] Sha BE, Onorato M, Bartlett JA, Bosch RJ, Aga E, Nokta M, Adams EM, Li XD, Eldridge J, Pollard RB. Safety and immunogenicity of a polyvalent peptide C4-V3 HIV vaccine in conjunction with IL-12. AIDS. 2004 May 21;18(8):1203-6. doi: 10.1097/00002030-200405210-00015. PMID 15166537
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067
- [Derived] Kalams SA, Parker S, Jin X, Elizaga M, Metch B, Wang M, Hural J, Lubeck M, Eldridge J, Cardinali M, Blattner WA, Sobieszczyk M, Suriyanon V, Kalichman A, Weiner DB, Baden LR; NIAID HIV Vaccine Trials Network. Safety and immunogenicity of an HIV-1 gag DNA vaccine with or without IL-12 and/or IL-15 plasmid cytokine adjuvant in healthy, HIV-1 uninfected adults. PLoS One. 2012;7(1):e29231. doi: 10.1371/journal.pone.0029231. Epub 2012 Jan 5. PMID 22242162